CLINICAL TRIAL: NCT01538368
Title: Magnetic Resonance Cholangio-pancreatography (MRCP) for Suspected Bilio-pancreatic Disease: Should the Endoscopist Take a Second Look?
Brief Title: Magnetic Resonance Cholangio-pancreatography (MRCP) for Suspected Bilio-pancreatic Disease
Status: Completed | Type: Observational
Sponsor: Deutsche Klinik fuer Diagnostik (Other)
Responsible Party: Principal Investigator, Till Wehrmann, Head, Divison of Gastroenterology, DKD Wiesbaden, Deutsche Klinik fuer Diagnostik
Other Study IDs: TWehrmann
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2012-02

CONDITIONS: Suspected Bilio-pancreatic Disease
Keywords: MRCP; ERCP; EUS; Image interpretation; MRCP findings; endoscopic intervention(s)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The interpretation of Magnetic Resonance Cholangio-pancreatography (MRCP)-findings is primarily performed by radiologists who only in some cases have experience with the interpretation of endoscopic retrograde cholangiopancreatography (ERCP)-images. It is unclear if MRCP-interpretation by the radiologist is sufficient to decide which additional endoscopic procedures might be necessary in an individual case or if an additional MRCP-interpretation by the endoscopist renders any clinical impact.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older who were referred for pancreato-biliary endoscopy to our unit based on actual MRCP-findings. In all cases MRCP should have been performed within 4 weeks prior admittance and a written radiological report as well as the digital images must be available.

Exclusion Criteria:

* Patients who had any endoscopic interventions in our institution before and also patients who underwent MRCP at our hospital were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: During 1/2007 until 12/2009 consecutive patients who were referred for dedicated endoscopic procedures regarding suspected alterations of the pancreato-biliary ductal system (nearly exclusively for EUS and/or ERCP) to our unit based on actual MRCP-findings were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Endoscopic management | 1 day
  Did the MRCP-interpretation by the gastroenterologist alter the scheduled endoscopic interventions ?

SECONDARY OUTCOMES:
MRCP-interpretation | 1 day
  Are there differences in the MRCP-interpreatation beween the radiologist and the gastroenterologist.